CLINICAL TRIAL: NCT01900509
Title: A Phase I Trial of Bendamustine in Combination With Clofarabine and Etoposide in Pediatric Patients With Relapsed or Refractory Hematologic Malignancies
Brief Title: Bendamustine Hydrochloride, Clofarabine, and Etoposide in Treating Younger Patients With Relapsed or Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BECHEM; TEVA ISS (Other: Teva Pharmaceuticals); NCI-2013-01148 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Acute Leukemia
Keywords: Childhood leukemia; Childhood lymphoma; Bendamustine
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; Clofarabine; Etoposide; etoposide phosphate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All participants who meet eligibility for this study will follow the same treatment regimen.
  INTERVENTIONS: bendamustine, clofarabine, etoposide (or etoposide phosphate), dexamethasone.
  Interventions: Drug: Bendamustine; Drug: Clofarabine; Drug: Etoposide; Drug: Etoposide phosphate; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bendamustine — Route of administration: intravenously (IV) over approximately 60 minutes, days 1-5.
  Other Names: Treanda(R); Bendamustine hydrochloride
Drug: Clofarabine — Route of administration: IV days 1-5.
  Other Names: Clolar(TM); Clofarex
Drug: Etoposide — Route of administration: IV days 1-5.
  Other Names: VP-16; Vepesid(R)
Drug: Etoposide phosphate — Route of administration: Used in substitution for etoposide in participants who experience allergic reaction, Etopophos® will be administered IV.
  Other Names: Etopophos(R)
Drug: Dexamethasone — Route of administration: three times daily orally (by mouth), days 1-5.
  Other Names: Decadron(R)

SUMMARY:
Participants with relapsed or refractory leukemia or lymphoma will be recruited for this study to find whether or not the addition of a new drug called bendamustine will be safe and possible to give with other chemotherapy drugs. This drug is approved by the Food and Drug Administration (FDA) for the treatment of other cancers in adults that are similar to those being studied in the research trial.

PRIMARY OBJECTIVES

* To establish the maximum tolerated dose (MTD) of bendamustine in combination with clofarabine and etoposide in pediatric participants with hematologic malignancies.
* To characterize the safety profile and dose-limiting toxicities (DLTs) of bendamustine in combination with clofarabine and etoposide.

SECONDARY OBJECTIVES

* To estimate event-free survival at 4 months.
* To estimate minimal residual disease (MRD) levels present at end of each cycle of therapy in participants with leukemia.
* To characterize the pharmacokinetic profile of bendamustine in the proposed regimen.

DETAILED DESCRIPTION:
Bendamustine will be combined with clofarabine and etoposide in a five-day cycle. Dexamethasone will be given to prevent capillary leak syndrome associated with clofarabine.

If the participant does not develop progressive disease or a dose-limiting toxicity (DLT) during the first cycle, a second cycle may be administered as a bridge to transplant. Each cycle lasts 21-28 days (or until count recovery).

Concomitant intrathecal therapy can be given at the investigator's discretion, but not on the same days as chemotherapy. Recommendations are triple intrathecal therapy (methotrexate, hydrocortisone, cytarabine) weekly for participants with CNS2 or CNS3 disease, and every two weeks for participants with CNS1 disease. Leucovorin may be given according to institutional guidelines.

The intent of this study design is for all participants to receive and complete one course of therapy. Participants who exhibit signs of disease progression or experience an unacceptable toxicity will be discontinued from protocol treatment.

ELIGIBILITY:
INCLUSION CRITERIA

* Participants with Hodgkin or Non-Hodgkin lymphoma must meet one of the following criteria: (a) Relapsing disease in 2nd or greater relapse and measurable disease, or (b) Refractory disease failing to achieve complete remission (CR) with > 2 induction or re-induction attempts.
* Participant with acute leukemia must meet one of the following criteria: (a) Relapsing acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML), or acute biphenotypic leukemia in 2nd or greater relapse; or (b) Refractory ALL, AML, or acute biphenotypic leukemia failing to achieve CR with ≥ 2 induction or re-induction attempts.
* Participant with leukemia has M2 or M3 marrow at the time of enrollment. Participant with M2 marrow must have definite cytogenetic, molecular, or immunophenotypic evidence of recurrent/refractory disease.
* Age is ≤ 21 years (participant has not yet reached 22nd birthday).
* Karnofsky or Lansky performance score is ≥ 60%. The Lansky performance score should be used for participants < 16 years and the Karnofsky performance score for participants ≥ 16 years.
* There are no known contra-indications to any of the planned agents used in this protocol. Etoposide may be substituted by etoposide phosphate (etopophos) if the patient has a history of hypersensitivity reaction to etoposide
* Adequate renal function defined as glomerular filtration rate > 60 cc/min/1.73m2, or normal serum creatinine based on age.
* Adequate hepatic function: (a) Direct bilirubin ≤ upper limit of normal (ULN) for age, or if total bilirubin is > ULN, direct bilirubin is ≤ 1.4 mg/dl, and (b) AST and ALT ≤ 5 x ULN for age.
* Adequate cardiac function defined as shortening fraction of ≥ 27% or ejection fraction ≥ 45%.
* Lymphoma participants without bone marrow involvement must have: (a) Absolute neutrophil count (ANC) ≥ 1,000/µL, and (b) Platelet count > 50,000/mm^3 (without transfusion support). [Note: these criteria are waived for participants with leukemia or lymphoma participants with bone marrow involvement.]
* Participant must have recovered from the acute side effects of all prior anti-cancer therapy, and :

  * At least 2 weeks have elapsed since prior systemic cytotoxic chemotherapy (except intrathecal chemotherapy, and/or low dose maintenance therapy such as vincristine, mercaptopurine, methotrexate or glucocorticoids), and
  * At least 4 weeks have elapsed since treatment with an investigational agent or antibody-based therapy, if applicable, and
  * If the participant received a prior allogeneic hematopoietic stem cell transplantation (HSCT), at least 3 months have elapsed and there is no evidence of active graft-versus-host disease (GVHD), participant has discontinued immunosuppression, and there is no history of veno-occlusive disease.

EXCLUSION CRITERIA

* Active, uncontrolled infection or severe concurrent medical disease, including but not limited to congestive heart failure, cardiac arrhythmias, or psychiatric illness.
* Isolated extramedullary disease (leukemia).
* Primary CNS lymphoma.
* Pregnant or lactating (female participant of childbearing potential must have negative serum or urine pregnancy test required within 7 days prior to start of treatment).
* Known HIV or active hepatitis B or C infection.
* Known hypersensitivity to bendamustine or mannitol.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Continually throughout the study (up to 3 months)
  Establish MTD of bendamustine in combination with clofarabine and etoposide.
Dose limiting toxicities | Continually throughout the study (up to 3 months)
  Characterize safety profile and DLTs of bendamustine in combination with clofarabine and etoposide

SECONDARY OUTCOMES:
Event free survival | 4 months after the start of therapy for the last patient enrolled on the study
  Event-free survival (EFS) time will be calculated from on therapy to any kind of failure or to last contact date for participants who are alive without any failure at the last contact date. The time to EFS will be set to 0 for participants who fail to achieve complete remission. Kaplan-Meier estimates of EFS curves will be computed, along with estimates of standard errors by the method of Peto. Four month EFS, as well as longer term survival rates (6 month and 1 year) will be estimated with 95% confidence intervals.
Proportion of leukemia participants with positive minimal residual disease | At end of each cycle of chemotherapy (approximately at 1 month and 2 months)
  The prevalence of MRD at end of each cycle is defined as proportion of MRD positives; we will estimate these proportions with point and interval estimates.
Plasma concentration of bendamustine | Day 1 and day 5 of cycle 1 therapy
  Plasma concentrations of bendamustine will be measured using an established LC-MS/MS assay. Bendamustine pharmacokinetic parameters such as Cmax, tmax, AUC (0-t), t1/2, and clearance will be estimated using population-based modeling techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Jeha S, Crews KR, Pei D, Peyton M, Panetta JC, Ribeiro RC, Zhao X, Campbell P, Metzger ML, Yang JJ, Cheng C, Pui CH, Bhojwani D. Phase 1 study of bendamustine in combination with clofarabine, etoposide, and dexamethasone in pediatric patients with relapsed or refractory hematologic malignancies. Cancer. 2021 Jun 15;127(12):2074-2082. doi: 10.1002/cncr.33465. Epub 2021 Feb 17. PMID 33598942
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols